CLINICAL TRIAL: NCT05905263
Title: The Effect of Virtual Reality Application on Student Satisfaction, Self-Confidence, and Anxiety Levels in Episiotomy Training
Brief Title: The Effect of Virtual Reality Application on Student Satisfaction, Self-Confidence, and Anxiety Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Demet Guney, MSc., Research Assist, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/112
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Virtual Reality; Episiotomy
Keywords: Virtual Reality; Educational; Self-Confidence; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application group with virtual reality (Experimental): Each student will be introduced to the materials to be used for virtual reality and will be informed about the application. After the introduction and information is given, the lens and pupil distances of the virtual reality glasses will be adjusted according to each student and students will be asked to wear them on their heads. Students will then be required to wear gloves. The application will be made one-on-one with each student. The application will be carried out sitting in the laboratory. If the student experiences symptoms such as dizziness and nausea during the application, the application will be terminated. If the student wants to continue the practice after listening, it will be continued. While the students are in the application, the interface will be introduced through the images projected to the computer simultaneously.
  Interventions: Other: Application group with virtual reality

INTERVENTIONS:
Other: Application group with virtual reality — Each student will be introduced to the materials to be used for virtual reality and will be informed about the application. After the introduction and information is given, the lens and pupil distances of the virtual reality glasses will be adjusted according to each student and students will be asked to wear them on their heads. Students will then be required to wear gloves. The application will be made one-on-one with each student. The application will be carried out sitting in the laboratory. If the student experiences symptoms such as dizziness and nausea during the application, the application will be terminated. If the student wants to continue the practice after listening, it will be continued. While the students are inside the application, the interface will be introduced through the images projected to the computer simultaneously.
  Other Names: Calf tongue group

SUMMARY:
The study aims to develop a virtual reality application for episiotomy training and to determine the effect of the virtual reality application on student satisfaction, self-confidence, and anxiety levels.

It was found that there should be a total of at least 102 students, 51 of whom are Virtual Reality practice groups (experimental) and 51 Dana Language practice groups (control), who meet the inclusion criteria. Considering the losses, it was decided to include 110 students in the study.We are collected usıng a Personal Informatıon form, Student Satisfaction and Self-Confidence in Learning, State and Trait Anxiety Inventory- STAI I-II

DETAILED DESCRIPTION:
The study aims to develop a virtual reality application for episiotomy training and to determine the effect of the virtual reality application on student satisfaction, self-confidence, and anxiety levels.

As one of the most common surgical procedures in vaginal delivery, episiotomy or perineotomy is an incision procedure performed in the perineum. Episiotomy is a surgical incision made in the bulbocavernosus muscle in the perineum during the second stage of labor (Yıldız Karaahmet & Yazıcı, 2016). Episiotomy is often performed to ensure the easy, quick, and safe delivery of the baby's head, to prevent fetal hypoxia, to shorten the active phase of labor, to prevent lacerations, to protect the anal sphincter, and to prevent perineal problems after delivery (Durmaz & Buğdaycı, 2013, Kartal et al., 2014).

ACOG recommends episiotomy in case of maternal or infant risk, such as perineal tears that may occur during vaginal delivery, to facilitate or expedite labor, and to restrict its use when not necessary (ACOG, 2006). The prevalence of episiotomy varies between countries. For example, its prevalence is 3.7% in Denmark and 75% in Cyprus (Blondel et al., 2016). In Turkey, the prevalence of episiotomy is reported to be 64-88% (Karaahmet & Yazıcı, 2016). Episiotomy can cause perineal pain, puerperal infection, postpartum hemorrhage, and dyspareunia later in life (Yang & Bai, 2021). Considering the complications of episiotomy, it is extremely important to perform episiotomy correctly, and only when necessary. It is therefore essential that midwives responsible for this practice acquire the necessary knowledge and skills (Aytekin et al., 2022).

In midwifery education, training is provided both theoretically and in clinical practice to put into practice and reinforce theoretical knowledge. While providing psychomotor development and professional socialization of students, it is also necessary to support standard education and clinical practice with simulation methods (Uyar Hazar & Gültekin, 2019). The training by simulation method seems to be often used to provide effective and high-quality midwifery skills (Bingöl et al., 2020). This training is conducted in laboratory environments with realistic scenarios in the form of performing practices (Cofey, 2015). Various simulation materials (sponge, calf's tongue, chicken breast, episiotomy model) have been used to improve the episiotomy skills of midwifery students (Aytekin et al., 2022). Another simulation method is training with Virtual Reality (VR) method. The virtual reality method helps training by providing an environment that allows students to experience scenarios and situations instead of imagining them (Çapa, 2004). Virtual reality environments offer students the opportunity of detailed observations with new visualization methods and an environment without physical obstacles. VR also provides a learning experience on a platform where they can interact and learn independently (Torres et al., 2015). In the literature review, there were no studies on the application of virtual reality in episiotomy training.

In this regard, the primary aim of this study is to develop a virtual reality application in episiotomy training, and the secondary aim is to determine the effect of this virtual reality application on student satisfaction, self-confidence, and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd year student of the Midwifery Department,
* Not having received episiotomy training,
* Volunteer to participate in the study.

Exclusion Criteria:

* Not voluntarily participating in the study,
* Dizziness, nausea, etc. during the application. symptom development.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning | Baseline
  In the sub-dimension of satisfaction with learning; Five items measuring satisfaction with the teaching method, variety of learning materials, facilitation, motivation, and the suitability of simulation in general, self-confidence sub-dimension; The content adequacy includes eight items: self-confidence, content requirement, skill development, available resources, and information on how to get help to solve clinical problems in simulation. Responses are scored on a five-point Likert system, ranging from 1 (strongly disagree) to 5 (strongly agree), and the total score varies between 13-65.
State and Trait Anxiety Inventory- STAI I-II | Baseline
  It is a Likert-type scale that measures state and trait anxiety levels separately with 20 questions. High scores indicate high anxiety levels, low scores indicate low anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniy Dınc Kaya, Ph.D, Principal Investigator — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD avalilable.

REFERENCES:
- [Background] Barjon K, Vadakekut ES, Mahdy H. Episiotomy. 2024 Oct 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK546675/ PMID 31536281
- [Background] Blondel B, Alexander S, Bjarnadottir RI, Gissler M, Langhoff-Roos J, Novak-Antolic Z, Prunet C, Zhang WH, Hindori-Mohangoo AD, Zeitlin J; Euro-Peristat Scientific Committee. Variations in rates of severe perineal tears and episiotomies in 20 European countries: a study based on routine national data in Euro-Peristat Project. Acta Obstet Gynecol Scand. 2016 Jul;95(7):746-54. doi: 10.1111/aogs.12894. Epub 2016 Apr 5. PMID 26958827
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Yang J, Bai H. Knowledge, attitude and experience of episiotomy practice among obstetricians and midwives: a cross-sectional study from China. BMJ Open. 2021 Apr 12;11(4):e043596. doi: 10.1136/bmjopen-2020-043596. PMID 33846148
- Available data/document: Clinical Study Report — https://clinicaltrials.gov/ProvidedDocs/58/NCT04444258/Prot_SAP_ICF_000.pdf — DEVELOPMENT AND USAGE OF VIRTUAL REALITY APPLICATION IN TEACHING FETAL DEVELOPMENT